CLINICAL TRIAL: NCT01665157
Title: A Randomized, Single-blinded, Comparative Study to Evaluate the Efficacy and the Acceptability of Low-residue Diet Package (Enimaclin®) as Diet Control Before Colonoscopy
Brief Title: Efficacy and Acceptability of Low-Residue Diet Package (Enimaclin®) as Diet Control Before Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NTUH201109018RD
Record Dates: First submitted 2012-02-27; First posted 2012-08-15 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Dietary Modification
Keywords: Diet Control before Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low-residue diet package (Enimaclin®) (Experimental): Low-residue diet package with normal amount 2L PEG-ELS
  Interventions: Dietary Supplement: Enimaclin®; Drug: 2L PEG-ELS
- Self-controlled diet (Placebo Comparator): Self-controlled diet with normal amount of 2L PEG-ELS
  Interventions: Other: Self-controlled diet; Drug: 2L PEG-ELS
- Low-residue diet (Enimaclin®) package (Experimental): Low-residue diet package with low volume 1.5L PEG-ELS
  Interventions: Dietary Supplement: Enimaclin®; Drug: low volume 1.5L PEG-ELS

INTERVENTIONS:
Dietary Supplement: Enimaclin® — Enimaclin Colomil ® (Glico Co., Japan Osaka)，a low-residue diet package for each meal.
  The duration of study is one day before colonoscopy.
  Other Names: Enimaclin Colomil ®,a low-residue diet package
  Arms: Low-residue diet (Enimaclin®) package; low-residue diet package (Enimaclin®)
Other: Self-controlled diet — Self-controlled low residue diet.
  Other Names: Self-controlled low residue diet.
  Arms: Self-controlled diet
Drug: 2L PEG-ELS — Normal volume of PEG-ELS
  Other Names: Taiwan name: Niflec powder
  Arms: Self-controlled diet; low-residue diet package (Enimaclin®)
Drug: low volume 1.5L PEG-ELS — Low volume PEG-ELS
  Other Names: Taiwan name: Niflec powder
  Arms: Low-residue diet (Enimaclin®) package

SUMMARY:
The purpose of this study is to evaluate the efficacy and the acceptability of low-residue diet package (Enimaclin®) as diet control before colonoscopy.

DETAILED DESCRIPTION:
In this study, we investigate a randomized, single-blinded, comparative study to evaluate the efficacy and the acceptability of low-residue diet package (Enimaclin®) as diet control before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Outpatient or healthy volunteer for health examination, 20~75 years old
* Eligible for oral bowel preparation
* BMI (Body Mass Index) ≤ 30

Exclusion Criteria:

* Patients with severe constipation (as fewer than three stools per week)
* Patients with bowel obstruction
* Patients contraindicated with treatment drug
* Patients who need emergency medication
* Ineligible for bowel preparation
* Pregnant or breast-feeding
* Patients with known allergies to treatment drug or low-residue diet package
* Patients who are ineligible to enroll

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo Chiu, M.D., Ph.D., Principal Investigator — NTUH
Locations (4):
- Taiwan (4):
  - E-Da Hospital, Kaohsiung, Taiwan
  - National Taiwan University Hospital Bei-Hu Branch, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Medical University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 14 months Recruitment location: GI outpatient clinic
Groups:
- Low-residue Diet Package and 2L PEG: Low-residue diet package (Enimaclin) with normal amount 2L PEG-ELS
- Self-controlled Diet and 2L PEG: Self-controlled diet with normal amount 2L PEG-ELS
- Low-residue Diet Package and 1.5L PEG-ELS: Low-residue diet package(Enimaclin) with low volume 1.5L PEG-ELS
Period: Overall Study
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package and 1.5L PEG-ELS
Started | 60 | 60 | 60
Completed | 60 | 60 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low-residue Diet Package (Enimaclin®) and 2L PEG: Low-residue diet package with normal amount of 2L PEG-ELS
- Self-controlled Diet and 2L PEG: Self-controlled diet with normal amount of 2L PEG-ELS
- Low-residue Diet (Enimaclin®) Package and 1.5L PEG: Low-residue diet package with normal amount of 1.5L PEG-ELS
- Total: Total of all reporting groups
Arm/Group | Low-residue Diet Package (Enimaclin®) and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet (Enimaclin®) Package and 1.5L PEG | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 49 | 54 | 157
  >=65 years | 6 | 11 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.6) | 51.3 (12.7) | 53.0 (11.0) | 52.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 24 | 81
  Male | 32 | 31 | 36 | 99
Region of Enrollment [Number; unit: participants]
  Taiwan | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Overall Cleansing Level at Colonoscopy by Ottawa Bowel Preparation Scale
Description: Ottawa preparation scale: Colon is defined into 3 segments: Right(cecum, ascending), mid(transverse, descending), rectosigmoid. Each is scored from 0 to 4, 0 is best and 4 is worst. Fluid quantity of whole is scored as 0, small; 1, moderate; 2 large amount. The scale will be summation of the clearness of 3 segments of colon and overall fluid quantity. It ranged from 0 to 14, 0 is the most clean colon and 14 is the most dirty one. Segment score will be analyzed separately as continuous variable.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low-residue Diet Package Plus 1.5L PEG: Low-residue diet package(Enimaclin) with low volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package Plus 1.5L PEG
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 2.58 (2.15) | 3.22 (3.08) | 2.97 (2.79)
Statistical Analysis 1: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG vs Low-residue Diet Package Plus 1.5L PEG; Test type: Superiority or Other; p = 0.435, ANOVA — Not significant

2. Primary Outcome: Overall Cleansing Level at Colonoscopy by Aronchick Scale
Description: The overall proportion of participants scored as Excellent or Good by Aronchick scale.
  Description of Aronchick scale:It categorized colon cleansing into 5 level: Excellent, good, fair, poor, inadequate. It is categorical and cannot be summed. We will present
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Groups:
- Low-residue Diet Package Plus 1.5L PEG-ELS: Low-residue diet package(Enimaclin) with reduced volume low volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package Plus 1.5L PEG-ELS
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants | 91.7 | 76.7 | 78.3
Statistical Analysis 1: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG vs Low-residue Diet Package Plus 1.5L PEG-ELS; Test type: Superiority or Other; p = 0.046, Chi-squared
Statistical Analysis 2: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG; Null hypothesis: "Low-residue diet package and 2L PEG" vs. "Self-controlled diet and 2L PEG" provides same preparation quality; Test type: Superiority or Other; p = 0.024, Chi-squared
Statistical Analysis 3: Comparison: Low-residue Diet Package and 2L PEG vs Low-residue Diet Package Plus 1.5L PEG-ELS; Test type: Superiority or Other; p = 0.041, Chi-squared

3. Secondary Outcome: Willingness to Choose the Same Protocol After Different Low Residual Diet and PEG-ELS Protocol
Description: It represent the proportion of participants who wanted to choose the same protocol as they received in this trial.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Groups:
- Low-residue Diet Package and 1.5L PEG: Low-residue diet package(Enimaclin) with low volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package and 1.5L PEG
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants | 93.3 | 90.0 | 95.0

4. Primary Outcome: Total Volume of Purgatives That Ingested
Description: The total volume of PEG-ELS (Liter) that ingested or could be ingested by examinee before colonoscopy
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package and 1.5L PEG
Number analyzed (Participants) | 60 | 60 | 60
Liter | 1.96 (0.16) | 1.98 (0.12) | 1.61 (0.27)

5. Secondary Outcome: Satisfaction of Different Low Residual Diet and Bowel Preparation Protocol
Description: It represented the percentage of participants who is satisfied with the protocol.
Time Frame: 1 day
Measure: Number; unit: Percentage of participants
Groups:
- Low-residue Diet Package and 1.5 L PEG-ELS: Low-residue diet package(Enimaclin) with low volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package and 1.5 L PEG-ELS
Number analyzed (Participants) | 60 | 60 | 60
Percentage of participants | 73.3 | 36.7 | 76.7
Statistical Analysis 1: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG vs Low-residue Diet Package and 1.5 L PEG-ELS; Test type: Superiority or Other; p < 0.01, Chi-squared

6. Secondary Outcome: Convenience of Different Low Residual Diet and Bowel Preparation Protocol
Description: It represented the percentage of participants who thinks the protocol is easy to use.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Groups:
- Self-controlled Diet and 2L PEG: Self-controlled diet with 2L PEG-ELS
- Low-residue Diet Package and 1.5L PEG: Low-residue diet package(Enimaclin) with reduced volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package and 1.5L PEG
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants | 88.3 | 76.7 | 93.3
Statistical Analysis 1: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG vs Low-residue Diet Package and 1.5L PEG; Test type: Superiority or Other; p < 0.01, Chi-squared

7. Primary Outcome: Segmental Cleansing Level at Colonoscopy (Right Segment Preparation Failure)
Description: Segmental score of Ottawa bowel preparation scale was analyzed. The proportion of "right segment" preparation failure, defined as segmental score as "3 poor" or "4 inadequate", was presented.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Low-residue Diet Package and 2L PEG | Self-controlled Diet and 2L PEG | Low-residue Diet Package Plus 1.5L PEG
Number analyzed (Participants) | 60 | 60 | 60
percentage of participants | 1.7 | 15.0 | 6.7
Statistical Analysis 1: Comparison: Low-residue Diet Package and 2L PEG vs Self-controlled Diet and 2L PEG vs Low-residue Diet Package Plus 1.5L PEG; Test type: Superiority or Other; p = 0.025, Chi-squared

ADVERSE EVENTS:
Groups:
- Low-residue Diet Package: Low-residue diet package (Enimaclin) with normal amount 2L PEG-ELS
- Self-controlled Diet: Self-controlled diet with normal amount 2L PEG-ELS
- Low-residue Diet Package Plus 1.5L PEG-ELS: Low-residue diet package(Enimaclin) with low volume 1.5L PEG-ELS
Arm/Group | Low-residue Diet Package | Self-controlled Diet | Low-residue Diet Package Plus 1.5L PEG-ELS
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 1/60 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-residue Diet Package (N=60) | Self-controlled Diet (N=60) | Low-residue Diet Package Plus 1.5L PEG-ELS (N=60)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild abdominal pain noted after bowel preparation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No